CLINICAL TRIAL: NCT06336239
Title: PrevaLence of Albuminuria in Patients With CARdiovascular Disease and Type 2 Diabetes Mellitus in China: a National Cross-sectional Study
Acronym: PLACARD
Status: Recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Chang sheng Ma, Director of Cardiology, Beijing Anzhen Hospital
Other Study IDs: KS2023097
Record Dates: First submitted 2023-12-27; First posted 2024-03-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cardiovascular Disease; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The association between Cardiovascular Disease (CVD) and Chronic Kidney Disease (CKD) is well established. Traditional risk factors for CVD and CKD are similar, with type 2 diabetes mellitus (T2DM) being the most prevalent risk factor. However, CKD is underdiagnosed and undertreated in patients with CVD. Further understanding of the combination of CKD in CVD patients is important to formulate prevention and treatment strategies for CVD patients and high-risk groups, reduce adverse events in CVD patients, and prevent progression of CKD to End Stage Renal Disease (ESRD).

DETAILED DESCRIPTION:
The PLACARD study will include approximately 3,000 patients presenting to the cardiology department with type 2 diabetes and cardiovascular disease. The aim of this study was to assess the prevalence of proteinuria (urinary ACR) in type 2 diabetic patients with different cardiovascular diseases, both inpatient and outpatient in the cardiology departments of secondary and tertiary hospitals in China. Participants will be recruited at 30 clinical centers for a period of six months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* Diagnosed T2DM combined with ≥1 CVD (hypertension, coronary heart disease, atrial fibrillation, heart failure);
* During the data collection period, they went to the outpatient clinic of the cardiology department of the research center, or received treatment in the cardiology department;
* Ability to self-sign informed consent (electronic /paper).

Exclusion Criteria:

* Pregnant or lactating women;
* Dialysis patients;
* Other diseases that lead to elevated albuminuria, such as severe infection, confirmed primary glomerular disease, etc.;

  . Malignant tumors being treated (surgery, chemotherapy, radiotherapy or targeted therapy);
* Cachexia (CSS score ≥ 5 points);
* Severe liver disease (Child- Pugh grade C) ;
* Participated in an interventional clinical trial in the past three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will adopt a stratified, multi-level, and multi-center strategy for continuous screening to enroll patients who meet all inclusion criteria and none of the exclusion criteria. During the enrollment period, the Clinical Coordinator will communicate with and invite all potential patients attending the selected inpatient wards or the designated outpatient physicians
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The prevalence of albuminuria | On the day of patients enrollment.
  To assess the prevalence of albuminuria in patients who are combined with type 2 diabetes mellitus and different cardiovascular diseases in inpatient and outpatient cardiology departments of secondary and tertiary hospitals in China.

SECONDARY OUTCOMES:
Lthe prevalence of microalbuminuria and macroalbuminuria evels of microalbuminuria and macroalbuminuria | On the day of patients enrollment.
  To evaluate the levels of microalbuminuria and macroalbuminuria of patients with type 2 diabetes mellitus (T2DM) in inpatients and outpatients cardiology departments;
The prevalence of microalbuminuria and macroalbuminuria | On the day of patients enrollment.
  To evaluate the prevalence of microalbuminuria and macroalbuminuria in patients with T2DM complicated with different cardiovascular diseases
To evaluate the related influence factors of albuminuria and the treatment patterns of CKD patients and non-CKD patients in cardiology departments; | On the day of patients enrollment.
  After outpatient patients receive feedback on their renal function tests, assess whether physicians prescribe new relevant medical orders by recording them. Evaluate the treatment patterns for CKD and non-CKD patients in the cardiology department.
Evaluate the management of patients with type 2 diabetes mellitus and cardiovascular disease across different levels of cardiology departments in hospitals. | On the day of patients enrollment.
  Collect clinical assessment data from patients (including test results and the frequency of these tests over the past year), and assess the management of patient-related risk factors and complications by physicians in hospitals of different levels based on the frequency of testing.

OTHER OUTCOMES:
Exploratory Objective | On the day of patients enrollment.
  To evaluate the prevalence of retinopathy in T2DM patients with different cardiovascular diseases attending inpatient and outpatient cardiology departments in secondary and tertiary hospitals in China.

CONTACTS AND LOCATIONS:
Overall Officials: Changsheng Ma, Doctor, Principal Investigator — Beijing Anzhen Hospital
Locations (27):
- China (27):
  - Beijing Sixth Hospital, Beijing, Beijing Municipality
  - Fangshan District First Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chinese PLA Army Characteristic Medical Center, Chongqing, Chongqing Municipality
  - Haidong City Second People's Hospital, Haidong, Gansu
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Ruyang County People's Hospita, Luoyang, Henan
  - Luoyang Sixth People's Hospita, Luoyang, Henan
  - Yongcheng People's Hospital, Yongcheng, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhangjiagang Sixth People's Hospital, Zhangjiagang, Jiangsu
  - Shenyang Ninth People's Hospital, Shenyang, Liaoning
  - Shenyang Tenth People's Hospital, Shenyang, Liaoning
  - Jining First People's Hospital, Jining, Shandong
  - Tai'an First People's Hospital, Tai’an, Shandong
  - Weihai Central Hospital, Weihai, Shandong
  - Jing'an District Central Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University Qingpu Branch, Shanghai, Shanghai Municipality
  - Qinyuan County People's Hospital, Changzhi, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, XI Ail, Shanxi
  - The Fifth People's Hospital of Sichuan Province, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Taizhou Central Hospital, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT06336239/Prot_000.pdf